CLINICAL TRIAL: NCT03202342
Title: Functional Magnetic Resonance Imaging of Human Hypothalamic Responses to Taste, Temperature and Glucose Sensing
Brief Title: fMRI of Hypothalamic Responses to Taste, Temperature and Glucose
Acronym: COLD-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1302
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — Water; Glucose; ethyl butyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Water/gluc/gluc+EB/EB/gluc+EB_cold (Experimental): First Water 22 C, then Glucose 22 C, then Glucose + Ethyl butyrate 22 C, then Ethyl butyrate 22 C and then Glucose + Ethyl butyrate 0 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Water/gluc+EB/gluc/gluc+EB_cold/EB (Experimental): First Water 22 C, then Glucose + Ethyl butyrate 22 C, then Glucose 22 C, then Glucose + Ethyl butyrate 0 C and then Ethyl butyrate 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc/water/EB/gluc+EB/glucose+EB_cold (Experimental): First Glucose 22 C, then Water 22 C, then Ethyl butyrate 22 C, then Glucose + Ethyl butyrate 22 C and then Glucose + Ethyl butyrate 0 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc/EB/water/gluc+EB_cold/gluc+EB (Experimental): First Glucose 22 C, then Ethyl butyrate 22 C, then Water 22 C, then Glucose + Ethyl butyrate 0 C and then Glucose + Ethyl butyrate 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- EB/Gluc/gluc+EB_cold/water/glucose+EB (Experimental): First Ethyl butyrate 22 C, then Glucose 22 C, then Glucose + Ethyl butyrate 0 C, then Water 22 C and then Glucose + Ethyl butyrate 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- EB/gluc+EB_cold/gluc/glucose+EB/water (Experimental): First Ethyl butyrate 22 C, then Glucose + Ethyl butyrate 0 C, then Glucose 22 C, then Glucose + Ethyl butyrate 22 C and then Water 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc+EB_cold/water/glucose+EB/glucose/EB (Experimental): First Glucose + Ethyl butyrate 22 C, then Water 22 C, then Glucose + Ethyl butyrate 0 C, then Glucose 22 C and then Ethyl butyrate 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc+EB_cold/glucose+EB/water/EB/glucose (Experimental): First Glucose + Ethyl butyrate 22 C, then Glucose + Ethyl butyrate 0 C, then Water 22 C, then Ethyl butyrate 22 C and then Glucose 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc+EB_cold/gluc+EB/EB/water/glucose (Experimental): First Glucose + Ethyl butyrate 0 C, then Glucose + Ethyl butyrate 22 C, then Ethyl butyrate 22 C, then Water 22 C and then Glucose 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C
- Gluc+EB_cold/EB/gluc+EB/glucose/water (Experimental): First Glucose + Ethyl butyrate 0 C, then Ethyl butyrate 22 C, then Glucose + Ethyl butyrate 22 C, then Glucose 22 C and then Water 22 C
  Interventions: Other: Water; Other: Glucose; Other: Ethyl butyrate; Other: Glucose + ethyl butyrate; Other: Glucose + ethyl butyrate 0 C

INTERVENTIONS:
Other: Water — Water, 300 ml, at room temperature
Other: Glucose — Water containing 50 g glucose, 300 ml, at room temperature
Other: Ethyl butyrate — Water containing ethyl butyrate (pineapple flavour) 300 ml, at room temperature
Other: Glucose + ethyl butyrate — Water containing 50 g glucose and ethyl butyrate (pineapple flavour) 300 ml, at room temperature
Other: Glucose + ethyl butyrate 0 C — Water containing 50 g glucose and ethyl butyrate (pineapple flavour) 300 ml, at 0 degrees centigrade

SUMMARY:
The study will consist of five occasions with one week in between. BOLD signal intensity of the hypothalamus will be measured using fMRI. Measurements will be done before and after drinking 300 ml plain water or water to which glucose and/or ethyl butyrate will be added.

DETAILED DESCRIPTION:
The hypothalamus is known to be important for control of feeding behaviour as well as the regulation of temperature. Functional magnetic resonance imaging (fMRI) is a non-invasive method, which detects transient haemodynamic changes in the brain, using blood oxygen level dependent (BOLD) signal differences.

In order to investigate the role of hypothalamic neural activity in response to taste, glucose and temperature, fMRI will be performed before, during and after ingestion of 300 ml plain water or water with added ethyl butyrate (pineapple flavour), added glucose or added ethyl butyrate plus glucose. All beverages will be consumed at 22 °C and the combination will also be drunk at 0 °C.

The study uses a randomised cross-over design in 16 healthy male subjects with a normal body weight. There will be an interval of at least one week between the five occasions.

BOLD signal intensity of the hypothalamus will be continuously measured for 21 minutes (5 minutes baseline, 4 minutes during drinking and 12 minutes after drinking).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 25 years
* BMI between 20 and 23 kg/m2
* Length between 170 and 190 centimetres

Exclusion Criteria:

* Diabetes or history of other disturbances of glucose metabolism (eg impaired glucose tolerance, hypoglycaemia).
* Any genetic or psychiatric disease (e.g. fragile X syndrome, major depression) affecting brain
* Any significant chronic disease
* Renal or hepatic disease
* Recent weight changes or attempts to lose weight (> 3 kg weight gain or loss, within the last 3 months)
* Smoking (current or last 6 months)
* Alcohol consumption of more than 21 units per week or use of recreational drugs at present or in the last year
* Recent blood donation (within the last 2 months)
* Recent participation in other biomedical research projects (within the last 3 months), participation in 3 or more biomedical research projects in one year
* Contra-indication to MRI scanning:

  * Claustrophobia
  * Pacemakers and defibrillators
  * Nerve stimulators
  * Intracranial clips
  * Intraorbital or intraocular metallic fragments
  * Cochlear implants
  * Ferromagnetic implants

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-10-30 (Actual)

PRIMARY OUTCOMES:
Determine hypothalamic function in response to taste, temperature and glucose sensing | Before (5 minutes) and after (12 minutes) drinking
  BOLD-signal intensity

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van der Grond, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Opstal AM, Hafkemeijer A, van den Berg-Huysmans AA, Hoeksma M, Blonk C, Pijl H, Rombouts SARB, van der Grond J. Brain activity and connectivity changes in response to glucose ingestion. Nutr Neurosci. 2020 Feb;23(2):110-117. doi: 10.1080/1028415X.2018.1477538. Epub 2018 May 27. PMID 29806553